CLINICAL TRIAL: NCT05884385
Title: Exploring the Effect of Pre-surgery Simulated Warm-up and Mental Visualisation in Reducing Musculoskeletal and Cognitive Demands Experienced by Surgeons Performing Robot-assisted Laparoscopic Surgery
Brief Title: Effect of Surgeon Warm-up and Mental Visualisation During Robot-assisted Laparoscopic Surgery
Acronym: MURALS2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lancaster University (Other)
Collaborators: East Lancashire Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Abdulwarith Shugaba, Principal Investigator (MD Student), Lancaster University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: DEV046
Record Dates: First submitted 2023-04-05; First posted 2023-06-01 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Cognitive Deficit in Attention; Musculoskeletal Strain; Fatigue; Surgery
Keywords: Robot-assisted Laparoscopic surgery; Warm up; Mental Visualisation
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Intervention Model Description: Surgeons will perform 3 surgical procedures under 3 randomized conditions: no intervention, simulated exercises, and mental visualization. EMG and EEG monitoring will be performed to collect data at predefined POIs. Condition 1 involves no changes to their regular robotic procedure, while Condition 2 has surgeons perform simulated tasks before surgery. In Condition 3, surgeons undergo mental training scripts before performing surgery, which involves guided mental visualization. The study aims to investigate the effects of these conditions on surgical performance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No intervention (No Intervention): Surgeons performing procedures under this condition will receive no intervention. They will perform the robotic procedure as they would normally on a day-to-day basis without any change. EMG and EEG monitoring will be performed by collecting data at the various predefined POIs.
- Simulated exercises (Experimental): When surgeons perform procedures under this condition they perform the initial theatre briefing prior to starting an operating list. They then perform 5 minutes of a preloaded simulated task on the robotic console. These tasks are designed to emulate fundamental skills required to perform robot-assisted laparoscopic surgery. They will then proceed to perform surgery as they normally do whilst undergoing EMG and EEG motoring, collecting data at the predefined POIs.
  Interventions: Other: Simulated exercises
- Mental Visualisation (Experimental): Mental training scripts based on the different surgical procedures performed by the different specialties were developed using the Mackay nodal model of mental practice(34). This involves breaking down a task into individual steps called nodal points with detailed instructions which also incorporate sensory cues to enhance the mental representation in the eye of participants' minds.
  On the day of surgery, surgeons performing the procedure under this condition will consent to patients for their robotic procedure and then proceed to perform the initial theatre briefing prior to starting am operating list.
  After this, surgeons will then perform 5 minutes of guided mental visualisation rather than self-produced imagery will be performed using the mental training scripts. They will then proceed to perform surgery as they normally do whilst undergoing EMG and EEG motoring, collecting data at the predefined POIs.
  Interventions: Other: Mental Visualisation

INTERVENTIONS:
Other: Simulated exercises — as detailed in arm description
  Arms: Simulated exercises
Other: Mental Visualisation — as detailed in arm description
  Arms: Mental Visualisation

SUMMARY:
Study Design - A Counterbalanced Study

Aims - To determine the effect of a) warm-up exercises and b) mental visualisation on the musculoskeletal demands and cognitive demands respectively during robot-assisted laparoscopic surgery.

Outcome Measures -

1. EMG measurements of frequency and amplitude across muscle fibres.
2. EEG measurements of peak alpha power, and alpha spindle duration and amplitude.

Study Participants and Eligibility - Surgeons who have certificates of completion of training (CCT) and performing surgical procedures using the minimally invasive techniques of RALS.

Planned Size of Sample - The investigators have chosen the higher value for our power calculation (an effect size of 0.24) which requires 10 surgeons per condition performing 1 - 2 operations for 80% power to detect a difference between conditions, at an alpha of 0.05.

Planned Study Period-Duration - Each surgeon will be required to participate in the study for approximately 3 - 4 weeks performing 3 surgical procedures and based on estimates that surgeons routinely perform an average of 1 robotic procedure per week it is anticipated the study will run for 6 months.

Research Question - Does structured simulated warm-up exercises prior to performing surgery improve surgeons' ergonomic awareness and maintain the low muscle fatigue impact associated with RALS? The investigators also hypothesize that mental imagery, inducing a flow state associated with overall cortical synchronisation could decrease cognitive demands experienced by surgeons and potentially mitigate against the cognitive fatigue surgeons experience whilst performing procedures.

DETAILED DESCRIPTION:
BACKGROUND There is an increased utilisation of minimally invasive surgery (MIS) by virtue of it being more beneficial to patients, however, an increase in musculoskeletal (MSK) demands is observed when the modality of standard laparoscopic (LS) techniques are used compared with robot-assisted laparoscopic techniques (RALS). Studies have further highlighted that RALS is significantly associated with decreased musculoskeletal demands for surgeons, including findings from our recent study exploring the demands of RALS and LS surgery (MURALS study - NCT04477746).

Although most studies additionally observe that surgeons experienced less cognitive demands with RALS, the MURALS study on the other hand found that the favourable MSK effects associated with RALS come with a "cost" of concomitantly increasing surgeons' attentional demands. This finding is associated with the design of the robotic console's viewing cart which has a binocular design displaying high-definition 3-dimensional images similar to virtual reality headsets, thereby requiring fusion of images from both eyes to produce clear images of the operating field through the process of stereopsis. Also, this design of the viewing cart additionally acts to isolate the visual senses and block out other distractions within the surgeon's visual field.

The modern technology of RALS, therefore, offers better ergonomic advantages which could protect surgeons from adverse MSK effects and potentially prolong their surgical careers. The consequent effect of this would be an increase in the years' surgeons remain in active duty thereby being able to operate and provide life-changing treatments to an additional number of patients over the span of their careers.

Warm-up exercises, such as aerobic or stretching exercises and performing simulated tasks, all represent types of interventions associated with improved task performance, decreased completion times, and reduced errors. Warm-up exercises are routinely practiced by athletes before competing and amongst musicians and dancers prior to performances which are complex psychomotor tasks requiring high cognitive function and coordinated motor skill. Similarly, surgeons performing fundamental surgical skills like suturing performed simulations on mobile devices or on surgical simulators prior to being assessed using validated global rating scales like the Kundhal or Reznick scale demonstrated improved task performance, also consistent with the findings in a systematic review on the effect of warm-up exercises on surgical performance.

Another simple and inexpensive tool utilised by athletes to enhance performance is mental visualisation or mental imagery which is the cognitive rehearsal of tasks in the absence of physical movements for the purpose of mental rehearsal, relaxation or goal-setting purposes. Whilst athletes experience a myriad of different mental states during task performance, this technique of mental imagery has been shown to improve optimal performance in athletes by inducing, a flow state - which is characterized by automatic information processing without conscious thinking by suppressing prefrontal cortex activity temporarily. There is also an association between mental imagery and an observed greater power of alpha waves especially associated with the parietal (somatosensory processes) and occipital (visual processes) cortex. Studies in neurophysiology have clearly established that the neuroplastic changes observed during mental visualisation are similar to those which occur when physically performing tasks, due to the fact that performed or imagined movements stimulate the same neurons, engaging comparable patterns of connectivity between cortical motor regions.

Mental imagery has also been studied amongst surgeons, using the mind as a simulator for prior rehearsal of steps involved in a procedure with consequent improved overall performance and enhanced motor skills observed when surgeons performed both simple or complex procedures. Mental visualisation could therefore potentially serve as a tool for offsetting the cognitive demands associated with RALS.

The time-pressured, demanding nature of surgeons' jobs together with the working time directive leaves a little amount of time for training in methods to alleviate the demands associated with performing surgery. Therefore, warm-up exercises and mental visualisation can serve as simple, readily available, and cost-effective ways through which surgeons can maintain lower MSK demands and lessen the cognitive demands associated with RALS surgeons.

The Rationale for Current Study The investigators hypothesise that structured simulated warm-up exercises prior to performing surgery aimed at improving surgeons' ergonomic awareness will maintain the low muscle impact of RALS.

The investigators also hypothesize that mental imagery, inducing a flow state associated with overall cortical synchronisation could decrease cognitive demands experienced by surgeons and potentially mitigate against the cognitive fatigue surgeons experience whilst performing procedures, as observed in athletes demonstrating high alpha event-related synchronization when performing tasks.

The aim of this proposed study is to investigate the effect of warm-up exercises and mental visualisation in mitigating against the cognitive demands associated with RALS whilst retaining the advantage of decreased muscle demands.

Study Objectives To determine the effect of a) warm-up exercises and b) mental visualisation on the musculoskeletal demands and cognitive demands respectively during robot-assisted laparoscopic surgery.

To address these aims, the investigators will subject surgeons to three types of conditions: no intervention, simulated exercises pre-surgery as a form of warm-up exercise, and mental visualisation. These will be administered to surgeons whilst using cutting-edge physiological and neuroscientific methods to establish the mechanisms and patterns of fatigue associated with robot-assisted laparoscopic surgery.

Study Design and Data Collection Methods Study Setting Surgeons will be invited to take part in the study from East Lancashire Hospitals NHS Trust through their trust email addresses. Interested surgeons will then provide written informed consent before participating in the study, then they will be provided with study identification numbers in a sequential manner. A randomisation process maintaining the basic principles of sequence generation, allocation concealment, and implementation will be carried out using GraphPad software. This will provide the sequence of how each surgeon will be subjected to the different study conditions.

To avoid any unnecessary burdens, prior to the day of the first surgery, surgeons will complete validated questionnaires. These will include one regarding general health conditions using SF36 Health questionnaire and one regarding physical activity level using the International Physical Activity Questionnaire (IPAQ). Surgeons' basic demographic characteristics will be recorded on the first day of surgery including; age, BMI, handedness, glove size, and years of experience.

As part of the standard process of consenting patients for surgery, the surgeons or a member of the research team will inform the patients about the decision and consent provided by their surgeon to participate in the research study i.e. to allow data collection on their surgeon.

Robotic surgical procedures based on the specialty (e.g., nephrectomies, bowel resections, hysterectomies, hepatectomies) will be used for data collection by fitting Surgeons with both EMG and EEG wireless devices. This study is being conducted in real-life surgeries and controlling for conditions between operations will be uniquely challenging, therefore any operations where complications result in the surgery taking beyond 50% of the mean average surgery time, to prevent this skewing the data toward an effect increased musculoskeletal and cognitive demands. Data already collected will be stored and if applicable, analysis to the point of exclusion will be carried out, Because the surgical procedures are different between specialties, predefined points of interest (POI) which are similar between the various surgical procedures will be used as points of interest for data recording. These points of recording provide discrete areas of comparison because, the skills and techniques used at these points are similar and are expected to provide similar challenges to the surgeons and they will include the dissection of vessels, mobilisation of organs, dissection of target tissues, and suturing.

Study Outcome Measures Measurement of musculoskeletal demands (EMG) Electromyography (EMG) will be used to determine the varying degrees of musculoskeletal demands experienced by surgeons in the different experimental conditions whilst performing surgery using RALS. This will be achieved using Surface EMG which is a non-invasive procedure that measures muscle activity by recording the electrical signals generated within muscle fibres during contractions. EMG has been used to assess MSK demands in different settings, in athletes, dentists, and in surgeons, more recently in our MURALS study.

EMG data will be collected for 180 seconds at the predefined POIs throughout the surgery. The changes in muscle electrical activity noted on EMG will be used as a marker of MSK demands. For example, a reduction in amplitude with a corresponding increase in frequency indicates fatigue being induced, as the muscle's recruitment has changed to deal with the demand. Monitoring with be performed using the Four muscle groups (Biceps, Deltoid, Trapezius, and latissimus dorsi muscles) frequently associated with increased MSK demands when surgery is performed using MIS techniques. Because RALS is performed by surgeons sitting at the console, with a brow- and arm-rest, this considerably lowers the workload on the lower limbs, therefore these will not be included to avoid any confounding factors.

EMG protocol. Surgeons will scrub up and place the robotic ports required to insert instruments into the body cavity where the surgery will be performed. They then dock the robot's instrument cart before un-scrubbing. Before they proceed to the robotic control console, surgeons will be fitted with wireless EMG sensors. This will be done following standard and established procedures, over the skin which overlies the bellies of the four muscles and parallel to the muscle's fibres having an inter-electrode distance of 20mm. The EMG data collection procedures will follow established protocols regarding site preparation and electrode placement, as well as data collection, processing, and normalisation. A wireless EMG system has been selected so that it is minimally invasive and does not impede a surgeon's movement with wires.

Measurement of cognitive demands (EEG) Electroencephalography (EEG) will be used to determine the varying degrees of cognitive demands surgeons in the different experimental conditions experience whilst performing surgery using RALS. EEG measures the ongoing electrical activity of the brain across the scalp (standard EEG) or within the brain matter (intracranial EEG) during a given task. The investigators will utilise a wireless standard EEG device, which is a non-invasive technique and provides physiological quantification of an individual's neurophysiological state in real-time, which can be linked to cognitive function. This approach removes reliance on subjective measures such as self-report or questionnaires. Different brain waves are captured by EEG which reflect neural oscillations occurring at different frequencies.

The alpha-band frequency (8- 13 Hz) which is associated with a relaxed wakefulness state, and decreases with concentration has predominantly been used in studies as a proxy to index cognitive fatigue, however, beta wave activity (frequency of 13 - 20 Hz) has also been noted to increase with alertness level and decrease during drowsiness.

Alpha waves have been used in studies to measure cognitive fatigue both in drivers, train operators, and for the first time in surgeons in our MURALS study. The alpha-wave activity is considered to reflect individual fatigue states and can be quantified in terms of their peak frequency, duration, and amplitude, giving rise to an individual's alpha signature. There is also a large precedent in the literature relating observed changes in alpha power to be specifically associated with visual attentional demands. High alpha power has been associated with 'idling' of the cortex, when the brain is not actively processing information, and a decrease in alpha power from baseline indicates a change from a resting to an activated brain state because the cortical modules in visual areas display a smaller degree of cooperation and are less synchronized as they maintain visual encoding and processing, relative to baseline.

Further analysis of EEG data to scrutinize the behaviour and trend of beta wave activity will serve to strengthen observed findings in the study.

EEG protocol. Whilst surgeons are having EMG electrodes fitted, a similar procedure will be completed for the wireless Enobio 8 5G wireless EEG device (Neuroelectrics, Cambridge, MA, USA). Surgeons will be fitted with an appropriate size EEG electrode cap and electrode gel applied onto the scalp using the wells on the EEG cap. This does not interfere with the surgeon's comfort and if a surgeon requires the electrode cap to be removed during a procedure due to any reason, this can be performed seamlessly within a minute and without breaching sterility. a member of the research team who in addition to being an investigator on this project, is a medically qualified surgical trainee familiar with the theatre environment will perform this by asking the surgeon to step aside from the operating table, the electrode cap removed from any position of their comfort and their surgical cap put back in place.

Electrodes will be placed over the cortex using the eight channels montage: Cz, Fz, P7, P8, P3, P4, O1, and O2, in accordance with the international 10-20 Montage system. Similar to the EMG data capture, EEG data will also be collected during data will be collected for 180 seconds at the predefined POIs throughout the surgery.

Statistics and Data Analysis Plan All collected data will be anonymised and transferred to Lancaster University for data analysis. Data analysis will be facilitated by a Senior Lecturer in Research Methods for the undergraduate and postgraduate degrees at the School of Sport and Exercise Sciences.

EMG data analysis. Using recommended normalisation, sampling, filtering, and smoothing techniques data will be analysed using EMG Works (Delsys Inc., Boston, MA, USA). Change in EMG variables, such as frequency and amplitude, across the three experimental conditions, can provide information on how muscle fibre recruitment has changed and thus, provide an insight into the effects of the various interventions on MSK demands surgeons' experience.

EEG data analysis. Data will be collected and analysed using ENOBIO NIC1.4 software (Neuroelectrics, Spain) using standard referencing, sampling, filtering, and smoothing techniques. The different peak alpha powers, and alpha spindle duration and amplitude, across the three experimental conditions, will be noted. These will provide crucial information about what the cognitive demands are associated with the different interventions.

Statistical analysis To determine differences in musculoskeletal demands associated with warm-up exercises and the effect of mental imagery on cognitive demands, a repeated measure one - way within group ANOVA will be used to analyse the EMG and EEG data respectively to aid in drawing meaningful conclusions for dissemination using various academic mediums (publications and conferences).

This study should further highlight the benefits of reduced musculoskeletal demands associated with RALS and develop a case for incorporating warm-up exercises and mental visualisation to mitigate against the demands associated with performing minimally invasive surgery.

Sampling technique Power calculation and Sample Size Determination The investigators have used an A priori power calculation to compute the required sample size using G*Power 3. Warm-up exercises are estimated to improve surgical performance evidenced by higher Reznick composite mean scores, with a warm-up score of 22.96 and without warm-up of 19.33, p-value of ≤ 0.001(33). This is similar to the effect in another study showing significant differences between the warm-up versus the non-warm-up groups noted in median scores, 28.5 and 19.25 respectively, p = 0.042. Therefore address the effect of warm-up on surgeons, effect size is predicted to be (Cohen's d) of 4.62 however pragmatically using a small effect size of 1.5, the investigators will require 4 surgeons in each of warm-up and without warm-up conditions (total 8) with each surgeon performing 1 - 2 operations during each condition.

Mental imagery improves surgical performance with an effect size of 0.24 as reported in a meta-analysis exploring the role of mental training in the acquisition of surgical skills. Significant correlation with mental imagery and performance (ranging from 0.47-0.80) were obtained using Objective Structured Assessment of Technical Skills (OSATS) performance scores, therefore will use data from the 10 surgeons per condition to study this effect.

The investigators have chosen the higher of these three values for our power calculation (an effect size of 0.24) which requires 10 surgeons per condition performing at least 1 procedure during each experimental condition, for 80% power to detect a difference between the conditions, at an alpha of 0.05.

The investigators aim to collect at least 10% additional data per surgeon to mitigate against factors which can affect data collected as previously noted in the previous similar study the investigators conducted in surgeons, for example procedures being converted to open surgery or missing data points due to equipment errors.

4.5 Participant/Sample Recruitment Surgeons: The investigators will screen between 10 - 15 surgeons, aiming to recruit at least 10, who have completed their surgical training and currently consultant grade surgeons in the National Health Service (NHS) from various specialties; Urology, Gynaecology, Hepato-pancreatic and Colorectal Surgery, which are specialties that perform procedures involving abdominal and pelvic organs, where the benefit of RALS has mainly been demonstrated.

This will be a counterbalanced design where surgeons will be subjected to all 3 conditions; no interventions performed, simulated exercise - performing pre-surgery warm up tasks, and mental imagery - performing pre-surgery mental visualisation. All surgeons will undergo the three conditions which will enable uniformity and facilitate meaningful comparisons between the study conditions.

Any procedures with complications or significant difficulty will be excluded as this could serve to confound the findings of the study.

Participant/Sample identification Prior informal information about the study will be disseminated during surgical departmental meetings and the Blackburn Research Innovation Development group in general surgery (BRIDGES) meetings. Email addresses of Surgeons will be identified from the various workforce managers of the surgical departments and Surgeons will be contacted via their trust emails and will be provided with a brief introduction to the study and the Participant information Sheet (PIS). Surgeons who meet the inclusion criteria and perform operations using RALS and have expressed interest in participating in the study will then be selected and have a meeting arranged for consenting onto the study.

During this meeting a member of the research team will go through the PIS in details and answer any queries raised and the EMG and EEG processes will be explained and how these fit into the surgeon's operation. Surgeons who decide to take part will be consented to the most current and up-to-date PIS and Informed consent form.

Based on the surgeon's diary and theatre lists, a day will be chosen when they have suitable operations (e.g., Bowel resection) to be performed via RALS and prior email reminder will be sent to confirm any changes to their general health, or presence of any musculoskeletal symptoms that may interfere with the study.

Subject coding will be carried out with sequential codes at the point of surgeons being recruited.

Participant Consent Process All surgeons participating in the study will be provided with research information packs describing the nature and goals of the research, and study consent form. This will also contain the contact details of members of the research team who will be available to clarify and answer any questions. Consent forms must be completed, signed, and dated after the surgeon has received detailed information about the study and made their decision. Consenting process will be carried out by any member of the study group.

As part of the consenting process, Surgeons will consent to verbally informing their patients that, they (the surgeons) are taking part in a research study and assure them the study will not in way affect their surgery and no data is being collected from them as patients. Research team members will also inform patients about this, especially when surgeons cannot facilitate due to clinical commitments or if the initial consent for surgery has already occurred. For patients being consented on the day of surgery, they will be informed about the study whilst being provided relevant information on their standard care in the day care unit by the surgeon or the research team.

No patient data is required hence, a patient consent will not be required for the study.

Consenting surgeons will have dates identified in their diaries when surgical procedures relevant to the study are selected. Surgeons are free to withdraw from the study without giving reasons and without prejudice at any time during the study.

Participant Withdrawal Criteria Any study participant may withdraw their participation at any time by contacting the CI or any members of the research. The surgeons will contact the PI or any member of the research team, who will note in the participant's record the date of the request together with the written notification of withdrawal of consent.

Study Interventions

The study involves each surgeon performing three surgical procedures under three different conditions:

Condition 1 - Surgeons will perform the robotic procedure as they would normally do without any changes. EMG and EEG monitoring will be conducted by collecting data at predefined POIs.

Condition 2 - Surgeons will perform a preloaded simulated task for 5 minutes on the robotic console that emulates fundamental skills required to perform robot-assisted laparoscopic surgery. They will then perform the surgery as they would normally do while undergoing EMG and EEG monitoring, collecting data at the predefined POIs.

Condition 3 - Mental training scripts based on the different surgical procedures will be developed using the Mackay nodal model of mental practice. Surgeons will perform 5 minutes of guided mental visualization using these scripts after performing the initial theatre briefing. They will then perform surgery as they would normally do while undergoing EMG and EEG monitoring, collecting data at the predefined POIs.

Overall, the study aims to investigate the impact of these three different conditions on the surgeons' performance during the surgical procedures, as measured by the EMG and EEG data collected at predefined POIs.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years (Adult participants)
* Surgeons who have acquired their certificate of completion of training (CCT)
* Surgeons with experience in performing procedures using RALS.

Exclusion Criteria:

* Surgeons with significant physical and musculoskeletal health conditions that would impede optimal performance of surgical procedures (e.g., severe arthritis, traumatic bony or soft tissue injuries)
* Surgeons with significant musculoskeletal pain or stiffness that would impede optimal performance of surgery.
* Surgeons with any cognitive symptoms like poor motor coordination, Loss of memory, visual disturbances, or headaches.
* Surgeons on any medications altering cognitive function like Psychoactive drugs, antidepressants and anticonvulsants

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Muscle demands | 20 weeks
  EMG measurements of Maximal Voluntary Contraction (MVC) changes across points of interest to establish the musculoskeletal demands of RALS.
Cognitive demands | 20 weeks
  EEG measurements of alpha activity during RALS to determine changes in cognitive demands.

CONTACTS AND LOCATIONS:
Locations (1):
- East Lancashire Hospitals NHS Trust, Blackburn, Lancashire, United Kingdom